CLINICAL TRIAL: NCT06519487
Title: Perceived Discrimination, Geography, and Demographic Effects on Immune Cell Function and Regulation
Brief Title: Social Experiences and Demographic Factors in the Regulation of Immune Cells
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morgan State University (Other)
Collaborators: Texas Christian University (Other); University of Maryland, Baltimore (Other); University of Baltimore (Unknown)
Responsible Party: Principal Investigator, Ingrid Tulloch, Associate Professor, Morgan State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2407001
Record Dates: First submitted 2024-07-18; First posted 2024-07-25 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Perceived Discrimination; RNA; Inflammatory Response
MeSH Terms: conditions — Perceived Discrimination

STUDY DESIGN:
Intervention Model Description: A crossover model is used to investigate whether geography, race, and ethnicity, interacting with laboratory discrimination conditions, affect immune cell function through genomic and epigenetic mechanisms, with perceived discrimination moderating the immune outcomes. Participants from each geographic region and belonging to one of three race or ethnic groups will experience race-based and non-race-based social exclusion and "washout" phases to mitigate carryover effects. For instance, participants might first experience race-based social exclusion, followed by an inclusion period (washout), and then non-race-based social exclusion, followed by another washout. Blood samples will be collected after each social exclusion to measure immune responses. Each participant will serve as their own control, facilitating within-subject comparisons to reduce variability due to individual differences, except on the variables of interest.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and the outcomes assessor will be blinded to the conditions to reduce bias. Participants will not be informed about the specific conditions (race-based exclusion or non-race-based exclusion) they are experiencing during Cyberball game and will be instructed not to discuss their experiences with the investigator or the outcomes assessor. All participant's questionnaire responses, blood, and saliva samples are labeled with anonymized codes (computer-generated ID numbers) to prevent identification of the condition order and Cyberball randomizes sequences automatically. The outcomes assessor, who will analyze the blood and saliva samples for immune cell function and genomic and epigenetic markers and the questionnaire, will be unaware of the participants' assigned conditions. Data analysis will be performed on de-identified datasets and randomization managed by a separate team member not involved in data collection or analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Mid-Atlantic: Non-Hispanic Black Order 1 (Experimental): Participants play Cyberball™ with virtual players who appear to be non-Hispanic White. The participant only receives the ball once during the entire game, while all the non-Hispanic White avatars will pass the ball back and forth with each other many times.
  After completing surveys and providing saliva and blood samples, participants play Cyberball, in which they receive the ball from virtual players an equal number of times as the other avatars, regardless of their ethnicity. During this round, participants play cyberball with virtual players who do not have any obvious ethnic differences from them. The participant again only receives the ball once during the entire game, while the other avatars that look similar to them pass the ball back and forth with each other a number of times. After completing surveys and providing blood samples, participants receive the ball from virtual players an equal number of times as the other avatars, regardless of their ethnicity.
  Interventions: Behavioral: Cyberball
- Mid-Atlantic: Non-Hispanic Black Order 2 (Active Comparator): Participants play Cyberball with virtual players who do not have any noticeable ethnic differences from them. The participants only receive the ball once during the entire game, but avatars that look similar to them pass the ball back and forth with each other several times. After completing surveys and providing saliva and blood samples, participants play Cyberball again but receive the ball from virtual players an equal number of times as the other avatars, regardless of the avatars' ethnicity. Participants play another session of Cyberball™ with virtual players who appear to be non-Hispanic White. The participant only receives the ball once during the entire game, while all the non-Hispanic White avatars will pass the ball back and forth with each other many times. After completing surveys and providing blood samples, participants again play Cyberball but receive the ball from virtual players an equal number of times as the other avatars, regardless of the avatars' ethnicity.
  Interventions: Behavioral: Cyberball
- Mid-Atlantic: Non-Hispanic White Order 1 (Experimental): Participants play Cyberball™ with virtual players who appear non-Hispanic Black, or Hispanic. The participant receives the ball once during the game, while all the non-Hispanic Black or Hispanic avatars will pass the ball back and forth with each other many times. After completing surveys and providing saliva and blood samples, participants play Cyberball, in which they receive the ball from virtual players an equal number of times as the other avatars, regardless of their ethnicity. During this round, participants play cyberball with virtual players who do not have any noticeable ethnic differences from them. The participant again only receives the ball once during the entire game, while the other avatars that look similar to them pass the ball back and forth several times. After completing surveys and providing blood samples, participants receive the ball from virtual players an equal number of times as the other avatars, regardless of their ethnicity.
  Interventions: Behavioral: Cyberball
- Mid-Atlantic: Non-Hispanic White Order 2 (Active Comparator): Participants play Cyberball with virtual players who do not have any noticeable ethnic differences from them. The participants only receive the ball once during the game, but avatars that look similar to them pass the ball back and forth with each other several times. After completing surveys and providing saliva and blood samples, participants play Cyberball again but receive the ball from virtual players an equal number of times as the other avatars, regardless of the avatars' ethnicity. Participants play another session of Cyberball with virtual players who appear to be non-Hispanic Black or Hispanic. The participant receives the ball once during the game, while all the non-Hispanic Black or Hispanic avatars will pass the ball back and forth with each other many times. After completing surveys and providing blood samples, participants again play Cyberball but receive the ball from virtual players an equal number of times as the other avatars, regardless of the avatars' ethnicity.
  Interventions: Behavioral: Cyberball
- Mid-Atlantic Hispanic Order 1 (Experimental): Participants play Cyberball™ with virtual players who appear to be non-Hispanic White. The participant receives the ball once during the game, while all the non-Hispanic White avatars will pass the ball back and forth with each other many times. After completing surveys and providing saliva and blood samples, participants play Cyberball, in which they receive the ball from virtual players an equal number of times as the other avatars, regardless of their ethnicity. During this round, participants play Cyberball with virtual players who do not have any noticeable ethnic differences from them. The participant again only receives the ball once during the entire game, while the other avatars that look similar to them pass the ball back and forth several times. After completing surveys and providing blood samples, participants receive the ball from virtual players an equal number of times as the other avatars, regardless of their ethnicity.
  Interventions: Behavioral: Cyberball
- Mid-Atlantic Hispanic Order 2 (Active Comparator): Participants play Cyberball with virtual players who do not have any noticeable ethnic differences from them. The participants only receive the ball once during the entire game, but avatars that look similar to them pass the ball back and forth with each other several times. After completing surveys and providing saliva and blood samples, participants play Cyberball again but receive the ball from virtual players an equal number of times as the other avatars, regardless of the avatars' ethnicity. Participants play another session of Cyberball™ with virtual players who appear to be non-Hispanic White. The participant only receives the ball once during the entire game, while all the non-Hispanic White avatars will pass the ball back and forth with each other many times. After completing surveys and providing blood samples, participants again play Cyberball but receive the ball from virtual players an equal number of times as the other avatars, regardless of the avatars' ethnicity.
  Interventions: Behavioral: Cyberball
- Southwest Non-Hispanic Black Order 1 (Experimental): Participants play Cyberball™ with virtual players who appear to be non-Hispanic White. The participant only receives the ball once during the entire game, while all the non-Hispanic White avatars will pass the ball back and forth with each other many times. After completing surveys and providing saliva and blood samples, participants play Cyberball, in which they receive the ball from virtual players an equal number of times as the other avatars, regardless of their ethnicity. During this round, participants play cyberball with virtual players who do not have any noticeable ethnic differences from them. The participant again only receives the ball once during the entire game, while the other avatars that look similar to them pass the ball back and forth several times. After completing surveys and providing blood samples, participants receive the ball from virtual players an equal number of times as the other avatars, regardless of their ethnicity.
  Interventions: Behavioral: Cyberball
- Southwest Non-Hispanic Black Order 2 (Active Comparator): Participants play Cyberball with virtual players who do not have any noticeable ethnic differences from them. The participants only receive the ball once during the entire game, but avatars that look similar to them pass the ball back and forth with each other several times. After completing surveys and providing saliva and blood samples, participants play Cyberball again but receive the ball from virtual players an equal number of times as the other avatars, regardless of the avatars' ethnicity. Participants play another session of Cyberball™ with virtual players who appear to be non-Hispanic White. The participant only receives the ball once during the entire game, while all the non-Hispanic White avatars will pass the ball back and forth with each other many times. After completing surveys and providing blood samples, participants again play Cyberball but receive the ball from virtual players an equal number of times as the other avatars, regardless of the avatars' ethnicity.
  Interventions: Behavioral: Cyberball
- Southwest Non-Hispanic White Order 1 (Experimental): Participants play Cyberball™ with virtual players who appear non-Hispanic Black or Hispanic. The participant receives the ball once during the game, while all the non-Hispanic Black or Hispanic avatars will pass the ball back and forth with each other many times. After completing surveys and providing saliva and blood samples, participants play Cyberball, in which they receive the ball from virtual players an equal number of times as the other avatars, regardless of their ethnicity. During this round, participants play cyberball with virtual players who do not have any noticeable ethnic differences from them. The participant again only receives the ball once during the entire game, while the other avatars that look similar to them pass the ball back and forth with each other several times. After completing surveys and providing blood samples, participants receive the ball from virtual players an equal number of times as the different avatars, regardless of ethnicity.
  Interventions: Behavioral: Cyberball
- Southwest Non-Hispanic White Order 2 (Active Comparator): Participants play Cyberball with virtual players who do not have any noticeable ethnic differences from them. The participants only receive the ball once during the entire game, but avatars that look similar to them pass the ball back and forth with each other several times. After completing surveys and providing saliva and blood samples, participants play Cyberball again but receive the ball from virtual players an equal number of times as the other avatars, regardless of their ethnicity. Participants play another session of Cyberball with virtual players who appear to be non-Hispanic Black or Hispanic. The participant only receives the ball once during the entire game, while all the non-white avatars will pass the ball back and forth with each other many times. After completing surveys and providing blood samples, participants again play Cyberball but receive the ball from virtual players an equal number of times as the other avatars, regardless of the avatars' ethnicity.
  Interventions: Behavioral: Cyberball
- Southwest Hispanic Order 1 (Experimental): Participants play Cyberball™ with virtual players who appear to be non-Hispanic White. The participant only receives the ball once during the entire game, while all the non-Hispanic White avatars will pass the ball back and forth with each other many times. After completing surveys and providing saliva and blood samples, participants play Cyberball, in which they receive the ball from virtual players an equal number of times as the other avatars, regardless of their ethnicity. During this round, participants play Cyberball with virtual players who do not have any noticeable ethnic differences from them. The participant again only receives the ball once during the entire game, while the other avatars that look similar to them pass the ball back and forth several times. After completing surveys and providing blood samples, participants receive the ball from virtual players an equal number of times as the other avatars, regardless of their ethnicity.
  Interventions: Behavioral: Cyberball
- Southwest Hispanic White Order 2 (Experimental): Participants play Cyberball with virtual players who do not have any noticeable ethnic differences from them. The participants only receive the ball once during the entire game, but avatars that look similar to them pass the ball back and forth with each other several times. After completing surveys and providing saliva and blood samples, participants play Cyberball again but receive the ball from virtual players an equal number of times as the other avatars, regardless of the avatars' ethnicity. Participants play another session of Cyberball™ with virtual players who appear to be non-Hispanic White. The participant receives the ball once during the game, while all the non-Hispanic White avatars will pass the ball back and forth with each other many times. After completing surveys and providing blood samples, participants again play Cyberball but receive the ball from virtual players an equal number of times as the other avatars, regardless of the avatars' ethnicity.
  Interventions: Behavioral: Cyberball

INTERVENTIONS:
Behavioral: Cyberball — Cyberball™ is a virtual social exclusion game that simulates social interactions and acute discrimination experiences in a controlled laboratory setting. The game involves passing a virtual ball between players represented by images. In this study, only the participant is a real player, while the other "players" are pre-programmed virtual avatars controlled by the experimenter using Cyberball software. The ethnicity of these virtual players can be manipulated by changing the stock photos used to represent them. Participants in the Race-Based Social Exclusion condition play Cyberball with virtual players who appear to be of a different ethnicity from the participant. In the Non-Race-Based Social Exclusion, the participant plays with virtual players who do not have any obvious ethnic differences from the participant, and social inclusion is a washout condition where the participant receives the ball from the virtual players, regardless of the ethnicity of the avatars.

SUMMARY:
Immune-mediated inflammatory diseases are a health burden for approximately seven percent of the population of Western nations. Preliminary data suggest variations in ethnic identity and/or geography influence discrimination experiences and inflammatory response trends. This study investigates how geography, ethnicity, and laboratory manipulation of discrimination experiences affect immune cell function and genomic regulation. Flow cytometry and immune cell stimulation will test monocytes collected from peripheral blood for functional effects. Next-generation transcriptomics and epigenomics will assess genomic and epigenetic mechanisms. The hypothesis is that geography, self-identified race, and ethnicity, interacting with laboratory discrimination conditions during the virtual ballgame Cyberball™, significantly affect immune cell function through genomic and epigenetic mechanisms, with perceived discrimination as a moderating factor on the immune outcomes. The transdisciplinary nature of the proposed study aims to provide valuable insights into differential susceptibility to immune-mediated inflammatory diseases across diverse populations. Uncovering these insights will better inform population-relevant interventions for immune-mediated inflammatory diseases.

DETAILED DESCRIPTION:
More than a third of the residents of the United States suffer from a chronic disease, with almost half involving dysregulated immune processes. Immune-mediated inflammatory diseases pose a public health burden in the United States. Preliminary data from previous work suggest that variations in ethnic identity and geography might influence discrimination experiences and inflammatory response trends. To investigate the functional implications of these findings, a multi-institutional study is proposed, examining how social experiences and demographic factors predict the regulation and activity of immune cells. Specifically, the hypothesis is that geography, self-identified race, and ethnicity, interacting with laboratory discrimination conditions, significantly affect immune cell function through genomic and epigenetic mechanisms, with perceived discrimination moderating the immune outcomes. Participants will provide saliva samples, complete psychosocial and demographic questionnaires, and play the virtual social exclusion game Cyberball™ in a randomly assigned block order. Acute discrimination experiences are manipulated by conditions during Cyberball. Virtual players, who appear to be of a different race from the participant, exclude them by not passing the participant the ball in the race-based exclusion condition. In the inclusion condition, the participant receives the ball regardless of participant and virtual player race. In the general social exclusion (not race-based), the players and participant races are similar to the inclusion condition, except that the participant does not receive the ball. The block of Cyberball and blood draws randomly assigned are either: 1) race-based social exclusion and inclusion first, a blood draw, then non-race-based social exclusion, inclusion, and blood draw, or 2) non-race-based social exclusion and inclusion, a blood draw and then the race-based social exclusion and inclusion and a blood draw. Baseline and post-first block inflammatory responses in saliva will be measured using enzyme-linked immunosorbent assays (ELISAs) to determine the concentration of cytokines like C-reactive protein, interleukin-6, and tumor necrosis factor-alpha. Flow cytometry and immune cell stimulation with toxin will test monocytes purified and sorted from the participant's blood for functional effects. Next-generation transcriptomics and epigenomics will assess differentially expressed RNA and methylation enrichment, emphasizing genes involved in inflammation signaling pathways. The data will be statistically analyzed using regression analysis and structural equation modeling to determine the relationship between discrimination, geography, immune cell function, and regulation while controlling for other socio-demographic factors. The findings could inform public health initiatives and interventions to reduce health disparities and improve outcomes for marginalized communities.

ELIGIBILITY:
Inclusion Criteria:

* Non-Hispanic Black, Non-Hispanic White, or Hispanic
* At least 18 years of age
* Lives within 25 miles of, works, or attends Morgan State University, The University of Baltimore or Texas Christian University

Exclusion Criteria:

* Anyone not identifying as either non-Hispanic Black, non-Hispanic White, or Hispanic,
* Under 18 years old
* Does not live within 25 miles of, works, or attends Morgan State University, the University of Baltimore or Texas Christian University

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2028-06-03 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Frequency of Perceived Discrimination Experiences | Survey response collected before the first Cyberball Sequence within 30 minutes of arriving at the lab) and score calculated during data analysis
  Before the game, participants will be asked to complete the "Everyday Discrimination Scale" designed to measure their perceptions of discrimination encountered in their everyday lives. This instrument prompts respondents to rate the frequency of discriminatory events in their daily lives, such as "being treated with less courtesy than others." Everyday Discrimination Scale Participants provide their responses on a scale that ranges from "0" for "never" to "5" for "almost every day." The summed responses provide a measure of how frequently they experienced discrimination. The summed score can range from 0 to 50; the higher the score, the more frequently participants perceived that they experienced discrimination. Additionally, participants specify whether these experiences are due to various factors, including race and gender.
Type, Timing and Frequency of Lifetime Discrimination Experiences | Survey response collected within 30 minutes after completing the first Cyberball Sequence and score calculated during data analysis]
  The "Experiences of Discrimination Scale" measures the type, timing, and frequency of discrimination. Participants answer "yes" or "no" to 9 types of unfair treatment, such as, "Have you ever been unfairly fired?" The sum of "yes" responses ranges from 0 to 9, with a score above 6 indicating many unfair treatments. Participants also specify if the unfair treatment was due to race, skin color, or other characteristics. The sum of responses related to ancestry, race, ethnicity, or skin color indicates the frequency of racial discrimination. Additionally, participants report the last time they experienced unfair treatment due to race or ethnicity, with responses from 1 ("past week") to 4 ("more than a year"). Lower scores indicate more recent occurrences.
Recent Discrimination and Perceived Ethnic Discrimination Score | Survey responses collected within 30 minutes after completing the Second Cyberball Sequence and score calculated during data analysis]
  The sum of response scores for the Recent Discrimination (a) and Ethnic Discrimination (b) subscale items of the "General Ethnic Discrimination Scale"provides the frequency of recent discrimination experience and includes a manipulation check for the validity of the recent Cyberball condition Recent Discrimination is calculated as the sum of responses to all (a) items ranging from a choice of 1 for "never" to 6 for "almost all the time. A summed minimum score of 18 corresponds to no lifetime discrimination, and a summed maximum score of 108 corresponds to the most frequent experience of perceived lifetime discrimination. Lifetime Discrimination is calculated as the sum of all (b) item responses ranging from a choice of 1 for "never" to 6 for "almost all the time. A summed minimum score of 18 corresponds to no lifetime discrimination, and a summed maximum score of 108 corresponds to the most frequent experience of perceived lifetime discrimination.
Recent and Lifetime Discrimination Stress Score | Survey responses collected within 30 minutes after completing the Second Cyberball Sequence and score calculated during data analysis
  The Cumulative response score from the Stress from Discrimination (c) items on the General Ethnic Discrimination Scale measures a person's perception of the stress of recent and lifetime unfair treatment due to a participant's racial/ethnic identity. Participants are asked to respond to the statement "How stressful was this for you?" for each discrimination experience. Response choices range from 1 for "not at all stressful" to 6 for "extremely stressful." Discrimination Stress is calculated as the sum of all (c) items on the General Ethnic Discrimination (GED) scale, where a summed score of 17 indicates little to no stress, and 102 indicates the highest amount of stress experienced due to recent and lifetime discrimination experiences.
Relationship between salivary and serum immune responses | Samples used in assay are saliva collected at baseline (30 mins before) and 40 minutes after the first Cyberball sequence, and serum is purified from whole blood collected 30 minutes after the first and second Cyberball sequence.
  Multiplex enzyme-linked immunosorbent assays (ELISA) will allow assessment of the pg/mL concentration of inflammatory cytokines in saliva and serum. These data will be used to calculate correlation coefficients that depict the magnitude and direction of the relationship between saliva and serum inflammatory cytokine concentration. The cytokines to be measured are Interleukin-1 beta (IL-1β), Interleukin-6 (IL-6), Tumor Necrosis Factor-alpha (TNF-α, and c-Reactive Protein (CRP).
Distribution and Quantity of Immune Cells in Whole blood | These data will be from whole blood samples collected 30 minutes after the first and 30 minutes after the second Cyberball sequence. The sequences are between 90 to 120 minutes apart separated by a washout period.
  To determine the quantity of each type of peripheral blood mononuclear cells (PBMCs) available after the different Cyberball sequences, the PBMCs will be sorted and quantified from whole blood collected 30 minutes after the first and 30 minutes after the second Cyberball sequence. A Sony SH800 cell sorter is used to perform Fluorescence-Activated Cell Sorting (FACS) with appropriate antibodies to identify T cells (CD3+), B cells (CD19+), NK cells (CD56+), and monocytes (CD14+CD16-, CD14+CD16+) and counts provided of viable cells with the cell counter.
Stimulated PBMC Cytokine Release | PMBCs purified from whole blood collected collected 30 minutes after the first and 30 minutes after the second Cyberball sequence are compared at 0, 2, 24 and 26 hours after incubation in LPS
  Cellular Cytokine release from (PBMCs) purified from the participant's whole blood is assessed in the presence or absence of stimulation with lipopolysaccharide (LPS) toxin. The LPS incubation time will vary in length, and ELISA will measure pg/ml concentration of IL-6, TNF-α, IL-1β, CRP
Gene expression levels | PMBCs purified from whole blood collected collected 30 minutes after the first and 30 minutes after the second Cyberball sequence
  RNA expression counts and distribution will be measured in PBMCs purified from participant whole blood collected participants after completing the first and second Cyberball sequences (collection tines separated by up 2 hours)

SECONDARY OUTCOMES:
Magnitude of Race/Ethnic Residential Segregation (Dissimilarity Index) | Questionnaire responses to the zip code items are collected within first 30 minutes in the lab and Index calculated during data analysis
  The Dissimilarity Index or DI measures Race/Ethnic Residential Segregation. We aim to measure the DI between non-Hispanic Black and non-Hispanic White, Hispanic and non-Hispanic White, and Hispanic and non-Hispanic Black populations. Census tract data from the participant's childhood zip code will be used to calculate the three childhood dissimilarity indices. The 2020 census tract data for the current zip code will be used in the equation for calculating this index. The equation for the index is DI=100×0.5× SUM(PxiPx-PyiPy) where Pxi and Pyi are the populations of groups x and y in census tract i, and Px and Py are the total populations of groups x and y in the overall geographic area. The DI ranges from 0 to 100, with scores less than 30 indicating low segregation, 30-60 indicating moderate segregation, and greater than 60 indicating high segregation.
Average Community Risk Protective Factors | Survey responses are collected within 30 minutes after completing the first Cyberball sequence and score calculated during data analysis
  "The Communities That Care Youth Survey" assesses Community risk and protective factors. Calculated average risk scores are based on responses to risk items, and calculated average protection scores are based on the protective items, with minimum and maximum average scores equaling 1 and 4, respectively.
  The average community risk is determined by calculating the average responses to items based on the five risk factors: Drug availability, norms for drug use, availability of handguns, neighborhood attachment, and community disorganization. A sample Community Risk item states:"If I wanted to get some marijuana, how easy would it be for me to get some?" response choices range from 1 for "Very hard to 4 for "Very easy." Average scores of less than 2 for the five factors indicate low community risk, and 3 or greater indicates high community risk.
Average Community Protective Factors | Survey responses are collected within 30 minutes after completing the first Cyberball sequence and score calculated during data analysis
  "The Communities That Care Youth Survey" assesses Community risk and protective factors. Calculated average protective factors scores are based on responses to protective items, with minimum and maximum average scores equaling 1 and 4, respectively.
  The Average Community Protection is determined by calculating the average responses to items on two protective factors: Opportunities and Rewards for prosocial involvement. A sample Community Protective item states: "My neighborhood offers lots of opportunities to participate in positive activities." With response choices ranging from 1 for "Strongly disagree" to 4 for "Strongly agree" Average scores lower than 2 indicate low community protection and a score of 3 or greater indicates high community protective factors.
Resilience | Survey responses are collected within 30 minutes after completing the second Cyberball sequence and the average response score calculated during data analysis
  The Brief Resilience Scale consists of six items that assess participants' resilience or buffer against stressful experiences. A sample item states, "I tend to bounce back quickly after hard times," with response choices ranging from 1 for "Strongly Disagree" to 5 for "Strongly Agree." The participant's Resilience Score is based on a calculated average of the response scores to the six items on the scale. The minimum possible average score is 1, and the maximum is 6. Scores below 3 indicate low resilience and scores above 4.31 indicate high resilience.
Frequency of recent stress | Survey responses are collected within 30 minutes after completing the first Cyberball sequence and Perceived Stress score calculated during data analysis
  The frequency of recent stress is calculated by summing the response scores on the ten-item "Perceived Stress Scale." The response options for each feeling or thought indicate the frequency with which it occurred, ranging from 0 for "Never" to 4 for "Very Often." Scores can be made by summing across all 10 items. Scores can range from 0 to 40, with higher scores indicating greater stress.
Degree of Morbidity | Survey responses are collected within 30 minutes after completing the second Cyberball sequence and the sum of response scores calculated during data analysis
  The sum of response items on the "Comorbidity Questionnaire" provides a single measure of the magnitude of chronic medical conditions faced by participants. The questionnaire can have up to fifteen items with twelve listed illnesses and options for participants to list an additional three items. One point if given each is given for the presence of the condition, with an additional point for receiving treatment for the condition, and another if the condition affects daily function.
  The Degree of Morbidity is calculated by summing the responses to the three components for each listed illness. The minimum score that can be earned is 0, and the maximum score is 45, with higher scores indicating greater morbidity.
Methylation Score | Methylsequencing of PMBCs purified from whole blood collected collected 30 minutes after the first and 30 minutes after the second Cyberball sequence
  The proportion of methylated to unmethylated cytosines at CpG sites around regulatory transcripts in the nuclear factor kappa-light-chain-enhancer of activated B cells (NF-κB) signaling pathway will be assessed in purified PBMCs

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Morgan State University, Baltimore, Maryland
  - Texas Christian University, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
The following de-identified data will be shared: self-report demographic and summary values of perceived psychosocial experiences, feelings, and health conditions from participant questionnaires; average concentration values for cytokines from saliva samples; count and average values of each mononuclear cell type from blood samples organized by discrimination condition; average cytokine concentration values released by immune cells purified from blood samples; RNA sequence counts, expression matrices, and dimensional analysis outcomes across cell types from mononuclear cells; percentage of methylation at individual CpG sites and average methylation levels in specific genomic regions from mononuclear cells; and the correlation coefficient between methylation and transcriptional data from mononuclear cells.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the end of the study period or as summary data are published in research reports (whichever comes first). The cleaned data files will be available at ) OpenICPSR or another field-specific repository listed at Repositories for Sharing Scientific Data to allow for management and sharing according to NIH guidelines and remain as long as allowed by NIH
Access Criteria: Deidentified data will be available by written permission.